# Exploring Enrollment and Engagement Trends in Individuals Managing Keratoconus: A Comprehensive Examination of Data on Keratoconus Clinical Trials

This document serves as the Informed Consent Form designed specifically for participants with keratoconus who are involved in the <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: February 23, 2024

Consent Document for Individuals in an Observational Research Initiative

Receiving an invitation to fill out this document suggests that you may be eligible to take part in an innovative observational clinical study targeting individuals grappling with keratoconus. This thorough guide outlines the primary objectives of the study, the research methodologies involved, and the potential outcomes, encompassing both positive and potentially adverse effects. Before deciding, it is crucial to comprehend fully the possible ramifications of your participation, and seeking advice from your healthcare provider can offer essential perspectives. If any part of this material raises questions or causes confusion, feel free to reach out to the researcher or the designated contact person.

Understanding the Importance of Clinical Trials in Managing Keratoconus

Keratoconus is a progressive eye condition characterized by the thinning and bulging of the cornea, the transparent front part of the eye. This structural change leads to a cone-like shape of the cornea instead of its normal round curvature. As a result, vision

becomes distorted, and individuals with keratoconus often experience astigmatism and nearsightedness.

The exact cause of keratoconus is not fully understood, but it is believed to involve a combination of genetic, environmental, and hormonal factors. It typically begins during the teenage years or early twenties and may progress over time.

Symptoms of keratoconus include blurred or distorted vision, increased sensitivity to light, and frequent changes in eyeglass or contact lens prescriptions. In the early stages, glasses or soft contact lenses may help manage the symptoms. As the condition progresses, special rigid gas-permeable contact lenses, or in severe cases, surgical interventions such as corneal cross-linking or corneal transplant, may be recommended.

Regular eye exams are crucial for detecting and managing keratoconus, allowing for early intervention to optimize visual outcomes.

Clinical trials dedicated to keratoconus play a pivotal role in assessing the safety and efficacy of innovative treatments crafted for this condition. They act as fundamental tools in determining whether new therapeutic options surpass existing modalities, offering substantial evidence for their broader adoption.

This study distinctly focuses on grasping the individual experiences of those confronting keratoconus, actively involved in a clinical trial that integrates medical interventions. The primary aim centers around a comprehensive examination of trial completion rates and voluntary withdrawals within this specific patient cohort.

# Engaging Actively in Clinical Trial Surveys

Your dynamic engagement holds immense significance in this observational clinical study, and we encourage you to openly share your thoughts and experiences. This involves completing questionnaires every two weeks, typically requiring 20-30 minutes of your time. Additionally, our team plans quarterly check-in calls to ensure ongoing support and your continued involvement in the trial.

It is crucial to emphasize that your participation in the survey component of this study is entirely voluntary. You can choose which questions to answer or complete the entire questionnaire based on your preferences. Moreover, you retain the freedom to withdraw

from the trial at any point. Recognizing the personal value of participating in a clinical study, we are committed to providing assistance while respecting your privacy.

Understanding the Importance of Observational Clinical Trials

Enrolling in this medical trial entails active participation in an observational study, a critical component of clinical research meticulously designed to glean insights through non-intrusive monitoring of patients adhering to their treatment protocols.

Researchers will solely observe your experience, comprehensively evaluating the outcomes of your condition without altering your treatment plan. This trial structure is vital for deepening our understanding of the inherent progression of a specific medical condition and its impact on individuals. Your voluntary involvement in this observational study substantially contributes to advancing medical knowledge and refining care for individuals with similar medical conditions.

Setting This Study Apart in the Landscape of Keratoconus Clinical Trials

Recognizing the distinctive features of this research study is imperative. It operates solely on an observational basis, indicating that your participation will not encompass specific therapies or interventions. To make an informed decision regarding potential participation in a clinical trial, understanding the spectrum of keratoconus clinical research, including interventional studies incorporating diverse treatment regimens, is crucial.

Making an informed decision about your potential involvement in a clinical trial demands an active approach, involving thorough research and comparison among trials. Resources such as ClinicalTrials.gov offer comprehensive information about <a href="keratoconus studies">keratoconus studies</a>. Furthermore, Power's specialized online platform presents a detailed catalog of ongoing <a href="keratoconus clinical trials">keratoconus clinical trials</a> actively seeking volunteers. Through meticulous exploration and a comprehensive understanding of various clinical trial categories, you can confidently decide whether or not to participate.

**Potential Advantages** 

While participants in this observational clinical research may not experience immediate benefits, their engagement holds the potential for substantial long-term impact. The data gathered from participants will play a pivotal role in shaping future strategies for involving individuals affected by keratoconus, potentially broadening the horizons of medical research. Those involved in this clinical trial have the capacity to ignite significant advancements in the field of medical research, potentially reshaping the landscape for future keratoconus patients.

### Possible Health Consequences and Risks

Comprehending potential health effects on participants, especially in studies evaluating new drugs, is crucial despite the progress made through clinical trials.

However, in observational clinical research, we employ a distinct approach to minimize these effects by refraining from administering experimental medications to participants. Our main emphasis remains on vigilant monitoring and evaluating outcomes, ensuring the prevention of any avoidable health risks.

### Safeguarding Your Privacy in the Research

Preserving the utmost confidentiality of your data stands as a central tenet of this study. To guarantee your anonymity, refrain from including any personal or identifiable information in your questionnaire responses. The dedicated research team is focused on enhancing privacy and security protocols. However, it is crucial to acknowledge that specific legal circumstances may necessitate the disclosure of personal data.

## **Exploring Diversity in Clinical Trials**

For those eager to delve into the intricate facets of diversity within clinical trials, a wealth of online resources awaits exploration.

Whether your goal is to grasp the complexities of challenges and opportunities associated with diversity in clinical trials or broaden your perspectives, the following resources can prove instrumental in this endeavor:

Boden-Albala, Bernadette, Salina P. Waddy, Noa Appleton, Heather Kuczynski, Emily Nangle, and Nina S. Parikh. "Recruitment, Inclusion, and Diversity in Clinical Trials." *The Science of Health Disparities Research* (2021): 413-428.

National Academies of Sciences, Engineering, and Medicine. "Strategies for ensuring diversity, inclusion, and meaningful participation in clinical trials: Proceedings of a workshop." (2016).

### **Participant Confirmation**

I affirm that I have dedicated the required time to comprehend and internalize the contents of the informed consent form, either through independent review or with the assistance of professionals who clarified its details. I am delighted to confirm that all my inquiries have been resolved to my satisfaction.

| Participant Name |
|-----------------------|
| Participant Signature |
| <br>Date |

### Facilitator's Verification

I affirm that I engaged in a comprehensive discussion with the participant, thoroughly explaining the intricacies outlined in this written document. My main aim was to guarantee the participant's complete understanding of the primary research objectives, the employed methodology, potential risks and benefits, and other crucial aspects of the keratoconus clinical trial.

| Printed Name of Assisting Researcher |
|--------------------------------------|
| Signature of Assisting Researcher |
| Date |